CLINICAL TRIAL: NCT00538057
Title: A Randomised, Double-blind, Placebo-controlled, Four-way Crossover Study to Compare the Pharmacodynamics and Pharmacokinetics of GW685698X and GW642444M When Administered Separately and in Combination as a Single Dose From a Novel Dry Powder Device in Healthy Subjects
Brief Title: Comparing Two Respiratory Drugs When Used In Combination And Separately From A Novel Inhaler Device In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HZA105871
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Healthy volunteers
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- arm 1 (Experimental): study drug
  Interventions: Drug: GW685698X & GW642444M

INTERVENTIONS:
Drug: GW685698X & GW642444M — study drug

SUMMARY:
A combination of the corticosteroid GW685698X and the long-acting ß2-agonist GW642444M is being developed for once daily administration for the maintenance treatment of asthma and COPD. GW642444M and GW685698X will be simultaneously co-administered from a single device and compared with GW642444M and GW685698X administered separately in order to determine whether co-administration affects the safety, tolerability, pharmacodynamic and/or pharmacokinetics of either compound.

ELIGIBILITY:
Inclusion criteria:

* Healthy adults aged between 18 and 60 years.
* Male subjects or female subjects of non child bearing potential.
* Body weight at least 50 kg and BMI within the range of 19-31 kg/m2 inclusive.
* No significant abnormality from ECG at screening.
* FEV1 at least 90% predicted and FEV1 / FVC ratio at least 0.7 at screening.
* Current non-smokers who have not used any tobacco products in the 12 month period preceding the screening visit and have a pack history of equal to or less than 5 pack years.

Exclusion criteria:

* Systolic blood pressure above 145 mmHg or a diastolic pressure above 85 mmHg unless the Investigator confirms that it is satisfactory for their age.
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
* Subjects who have suffered an upper or lower respiratory tract infection within 4 weeks of the screening visit.
* Liver function tests (AST, ALT or ALP) greater than 1.5 of the upper limit of laboratory reference range.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
* History of milk protein allergy.
* The subject has taken prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is the longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has taken oral corticosteroids less than 8 weeks before the screening visit
* The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit
* History of alcohol/drug abuse or dependence within 12 months of the study.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has donated a unit (450mL) of blood within the previous 16 weeks or intends to donate within 16 weeks after completing the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has tested positive for HIV antibodies.
* The subject has a positive pre-study urine drug screen.
* Positive CO or alcohol breath test at screening or on admission to the Unit.
* History of any adverse reaction including immediate or delayed hypersensitivity to any ICS, ß2-agonist or sympathomimetic drug. gefitinib or erlotinib) is permitted. Use of bevacizumab must have ended at least 40 days prior to date of first dose of study drug.
* Any anti-cancer therapy (surgery, tumor embolization, chemotherapy, radiation therapy, immunotherapy, biological therapy, or hormonal therapy) currently or within 14 days prior to date of first dose of study drug.
* Any ongoing toxicity from prior anti-cancer therapy that is greater than Grade 1 and/or that is progressing in severity.
* Known immediate or delayed hypersensitivity reaction or idiosyncracy to drugs chemically related to pazopanib.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-10-02 (Actual); Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-01 (Actual)

PRIMARY OUTCOMES:
Maximum heart rate | over 4 hours after dosing.
Blood pressure | changes over 12 hours.
Electrocardiogram | changes over 12 hours.
Change in peak expiry flow rate | changes over 24 hours.
Change in serum cortisol concentration | changes over 24 hours.

SECONDARY OUTCOMES:
Change in plasma drug concentration (AUC, Cmax, t1/2, tmax) | over 48 hours after dosing.
Change in blood potassium levels | within 4 hours of drug dosing.
Mean heart rate | over 4 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- [Derived] Kempsford R, Allen A, Bareille P, Hamilton M, Cheesbrough A. The pharmacodynamics, pharmacokinetics, safety and tolerability of inhaled fluticasone furoate and vilanterol administered alone or simultaneously as fluticasone furoate/vilanterol. Clin Pharmacol Drug Dev. 2015 Jan;4(1):2-11. doi: 10.1002/cpdd.160. Epub 2014 Dec 5. PMID 27127998
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study HZA105871 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/HZA105871?search=study&search_terms=HZA105871#rs
- Available data/document: Informed Consent Form: HZA105871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HZA105871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HZA105871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HZA105871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HZA105871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HZA105871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HZA105871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register